CLINICAL TRIAL: NCT07079410
Title: A Single-Arm, Prospective Phase II Clinical Study on the Neoadjuvant Sintilimab Plus Cetuximab in Locally Advanced Oral and Oropharyngeal Squamous Cell Carcinoma
Brief Title: Neoadjuvant and Adjuvant Sintilimab Plus Cetuximab in Locally Advanced Oral and Oropharyngeal Squamous Cell Carcinoma
Acronym: OSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-287R
Record Dates: First submitted 2025-07-04; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC); Oropharyngeal Squamous Cell Carcinoma; Resectable Oral and Oropharyngeal Squamous Cell Carcinoma
Keywords: locally advanced OSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Treatment + Surgery + Adjuvant Treatment (Experimental): Neoadjuvant Treatment + Surgery + Adjuvant Treatment Neoadjuvant treatment: The participants will receive 2 cycles of combination therapy (Sintilimab, Cetuximab). surgery: Primary tumor resection and/or lymph node dissection surgery 3 weeks from cycle 2 day 1. Adjuvant treatment: 3-8 weeks post-surgery and up to a total of one year. The participants will receive Sintilimab (q3w) therapy. Interventions: Drug: Sintilimab, Cetuximab
  Interventions: Drug: Sintilimab+Cetuximab

INTERVENTIONS:
Drug: Sintilimab+Cetuximab — Neoadjuvant treatment: the participants will receive Sintilimab 200 mg (each 3-week/cycle) and Cetuximab (400 mg/m2 first time and followed 250 mg/m2, day 1, day 8, day 15) for 2 cycles. Adjuvant treatment: the participants will receive Sintilimab 200 mg (each 3-week cycle, a total of 17 cycle) for a total of one year.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the combination therapy of immunotherapy (Sintilimab) with targeted therapy (Cetuximab) as a possible treatment before and after surgery for locally advanced oral/pharyngeal squamous cell carcinoma.

DETAILED DESCRIPTION:
Approximately 60% of patients with oral/oropharyngeal squamous cell carcinoma (OSCC) are found to be in the local advanced stage. Even if they actively undergo comprehensive sequential treatment such as surgery, radiotherapy, and chemotherapy, the 5-year survival rate is still less than 50%. According to both the NCCN and the CSCO head and neck cancer treatment guidelines, radical surgery is the main treatment strategy for locally advanced OSCC, and adjuvant radiotherapy or chemotherapy/radiotherapy. However, the high treatment failure rate and disease recurrence rate are still the fundamental reasons for its poor prognosis. In recent years, neoadjuvant therapy has been proven to reduce the burden of local diseases in multiple tumor types, thereby improving surgical outcomes, reducing the risk of distant metastasis, and predicting prognosis based on the patient's pathological response. The combination of anti-PD-1/PD-L1 monoclonal antibody and EGFR monoclonal antibody has a synergistic anti-tumor effect. Multiple prospective studies have shown that the combination of cetuximab and anti-PD-1 monoclonal antibody has achieved good efficacy in the treatment of recurrent/metastatic head and neck squamous cell carcinoma. The combination of neoadjuvant immunotherapy and EGFR monoclonal antibody therapy for locally advanced OSCC is worth exploring. This prospective, open label, single arm, phase II single center interventional study aims to evaluate the efficacy and safety of the neoadjuvant and adjunvant combination therapy of Sintilimab (anti-PD-1 monoclonal antibody) and cetuximab in patients with locally advanced OSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed oral/oropharyngeal squamous cell carcinoma (including tongue, lips, gums, cheeks, floor of mouth, hard palate, soft palate, posterior molar area, lateral pharyngeal wall, posterior pharyngeal wall, tonsils). PD-L1 expression score (CPS score) >1
2. Participants must diagnosed with clinical staging III or IVa (AJCC, 8th edition), without evidence of distant metastasis (M0) based on PET/CT or chest, abdominal and pelvic CT scans, and standard treatment is recommended, including surgical resection and adjuvant radiotherapy+/- chemotherapy.
3. Age ranges from 18 to 75 years old
4. ECOG performance status 0 or 1.
5. Expected survival ≥ 3 months.
6. Participants must have not received treatment for before.
7. There must be at least one clinically assessable lesion according to the RECIST V1.1 criteria prior to treatment.
8. The participants may have any human papillomavirus (HPV) status of the tumor. Patients with oropharyngeal cancer need to undergo HPV testing, including p16 immunohistochemistry and/or confirmatory HPV polymerase chain reaction (PCR) or in situ hybridization (ISH) testing.
9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and continue contraception for 12 months after the end of treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Participants must have adequate organ and marrow function as defined below: The function of important organs meets the following requirements: (1) normal bone marrow reserve function, white blood cell (WBC) ≥ 3.0 × 10 ^ 9/L; Neutrophil count (NEUT) ≥ 1.5 × 10 ^ 9/L, platelet count (PLT) ≥ 100 × 10 ^ 9/L, hemoglobin (Hb) ≥ 90 g/L; (2) Normal renal function or serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥ 50 ml/min (Cockcroft Gault formula); (3) Normal liver function or total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); AST or ALT levels ≤ 3 times the upper limit of normal (ULN); (4) Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously. If FT3 and FT4 levels are normal, they can be included in the group).
11. The participants voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Squamous cell carcinoma with primary site of nasopharynx or skin.
2. Diagnosed with malignant diseases other than head and neck squamous cell carcinoma within 3 years before the first administration (excluding Radical treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curative excised carcinoma in situ)
3. Has received therapy treatment with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, or anti-CTLA-4 antibody (or any other antibody acting on T cell co stimulatory or checkpoint pathways).
4. Has received live or attenuated vaccines within 30 days prior to the first dose of Sintilimab, inactivated vaccines are allowed.
5. Has received immunosuppressive drugs within 14 days prior to the first dose of study drug, nasal and inhaled corticosteroids or physiological doses of systemic corticosteroids (i.e. not exceeding 10 mg/day of prednisolone or other corticosteroids of equivalent physiological doses) are allowed.
6. Has an active infection that requires systematic treatment; Has a history of non -infectious pneumonia/interstitial lung disease requiring steroid treatment, or current pneumonia/interstitial lung disease; Has a known history of hepatitis B (defined as positive for hepatitis B surface antigen [HBsAg]) or known history of active hepatitis C virus (defined as detection of HCV RNA [qualitative]) infection; Has a known history of human immunodeficiency virus (HIV) infection.
7. Has received allogeneic tissue/solid organ transplantation.
8. Has not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 2) with the exception of alopecia.
9. Has obvious cardiovascular abnormalities (such as myocardial infarction, superior vena cava syndrome, and heart disease grade 2 or above diagnosed according to the New York Heart Association (NYHA) classification criteria within 3 months prior to the enrollment)。
10. Has severe clinical infection (>NCI-CTCAE 5.0 Level 2 infection);
11. Has uncontrollable hypertension (systolic blood pressure>150mmHg and/or diastolic blood pressure>90mmHg after treatment with antihypertensive drugs) or clinically significant cardiovascular diseases - such as cerebrovascular accidents (≤ 6 months before enrollment), myocardial infarction (≤ 6 months before enrollment), unstable angina, congestive heart failure classified as Grade II or above by the New York Heart Association (NYHA), or severe arrhythmias that cannot be controlled with medication or have potential impact on experimental treatment.
12. Pregnant women are not allowed to participate. Breast-feeding women who participate in this study should stop breast-feeding.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Has participated in other clinical studies within 30 days prior to enrollment.
15. Other situations that researchers consider unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Pathological Response (mPR) | 2 months
  Major pathologic response (mPR) is defined as having ≤ 10% invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes as assessed by pathologists. Rate is the proportion of treated participants who experienced mPR

SECONDARY OUTCOMES:
Rate of Pathologic complete response (pCR) | 2 months
  Pathologic complete response (PCR) is defined as having no invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes as assessed by pathologists. Rate is the proportion of treated participants who experienced PCR.
2 year Event-free Survival (EFS) Rate | 24 months
  EFS is the time from the date of study entry to the date of first record of disease progression as defined by RECIST 1.1
2 year Overall Survival (OS) Rate | 24 months
  OS is the time from study entry to death due to any cause
Adverse Events (AEs) | 24 months
  Number of participants experiencing any sign, symptom, disease, or worsening of preexisting conditions temporally associated with the experimental interventions or irrespective of the experimental interventions

OTHER OUTCOMES:
Changes in the Level of biomarkers for predicting therapeutic efficacy | 24 months
  Changes in the Level of PD-L1 expression, tumor mutation burden, microsatellite instability, immune cell invasion

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No